CLINICAL TRIAL: NCT03771300
Title: Efficacy of a Mindfulness-based Intervention Programme With or Without Virtual Reality Support to Reduce Stress in University Students: Protocol for a Randomized Controlled Trial
Brief Title: Efficacy of a MBI Programme With or Without Virtual Reality Support to Reduce Stress in University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Javier Garcia Campayo (Other)
Responsible Party: Sponsor-Investigator, Javier Garcia Campayo, Principal investigator, Hospital Miguel Servet
Organization: Hospital Miguel Servet (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FPU15/00598
Record Dates: First submitted 2018-12-02; First posted 2018-12-11 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Mental Health Wellness 1
Keywords: Wellness; University students; Mindfulness; Virtual Reality (VR)
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, pragmatic trial, involving three assessment time points (baseline, post-intervention and six-month follow-up).
Who Masked: Participant, Outcomes Assessor
Masking Description: The assignation of the subjects will be carried out after the evaluation by a member of the research group, who has no knowledge about the study, through a random sequence generated by computer. Participants will be assigned to one of these conditions: 1) Mindfulness condition; 2) Mindfulness condition complemented by VR environments; 3) Relaxation condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness condition (Experimental): 90-minute group sessions, held once a week over a space of 6 weeks, and is offered as an extra-curricular activity.
  Interventions: Behavioral: Mindfulness
- Mindfulness condition complemented by VR (Experimental): This condition is equivalent to the mindfulness condition (group sessions, held once a week over a space of 6 weeks and offered as an extra-curricular activity), unlike the time of each session, which is reduced from 90 to 75 minutes of duration.
  Interventions: Behavioral: Mindfulness condition complemented by VR
- Relaxation condition (Active Comparator): 90-minute group sessions, held once a week over a space of 6 weeks, and will be offered as an extra-curricular activity.
  Interventions: Behavioral: Relaxation

INTERVENTIONS:
Behavioral: Mindfulness — This program is structured around two central elements, mindfulness and compassion. The sessions combine theory and practice components, using a methodology which priorities the reflection and debate among the students. Regarding theory component, mindfulness and compassion concepts will be set out over the length of the program, in addition to others related to time management, stress, anxiety and the balance between personal life and academic/work life. The practical component of the program consists of mindfulness and self-compassion formal and informal practices under the guidance of a specialized instructor.
  Arms: Mindfulness condition
Behavioral: Mindfulness condition complemented by VR — The VR is comprised of a Samsung VR goggles, a Samsung Galaxy S6 phone and optional headphones.
  In this condition, the instructor is the same as previously but the implementation of VR will be carried out by a psychologist specially trained for the application of these VR scenarios. Prior to the VR use, the psychologist will make sure about the participants´ health.
  Arms: Mindfulness condition complemented by VR
Behavioral: Relaxation — This condition is based on the Progressive Muscle Relaxation.The relaxation program include training 16 muscle groups during the initial sessions, 7 muscle groups during the intermediate sessions, 4 muscle groups later and a only recall relaxation in the final session.This program is complemented with visualizations, as it was originally proposed by Jacobson (1938).
  Arms: Relaxation condition

SUMMARY:
There is a growing concern about mental health problems of university students. Stress, anxiety, and depression are reported to be common in this population. For this reason, mindfulness training is becoming increasingly popular in university contexts. This randomized controlled trial (RCT) pretends to evaluate the efficacy of a mindfulness-based intervention (MBI) to reduce levels of perceived stress and to improve the psychological well-being of university students. Besides, in response to the interest of young people for new technologies, this trial also pretends to explore the capacity of Virtual Reality (VR) to help adherence to the programme.

This study protocol presents an RCT, involving the assessment time points of baseline, post-intervention and six-month follow-up. A total of 280 students of the University of Zaragoza or National Distance Education University (UNED), in Spain, will be randomized to joining a mindfulness condition, a mindfulness condition complemented by VR environments, or a relaxation condition (active control group). Perceived stress will be the main outcome and will be measured using the 10-item self-report Perceived Stress Scale (PSS). Other well-being and academic functioning outcomes will also be assessed, as well as variables to explore the impact of VR. Multilevel mixed-effects models will be calculated to estimate the efficacy of the programme, and effect size estimations will be carried out. Effects of VR in adherence to the programme will be evaluated.

Some strengths of this study are the RCT study design, which includes a suitable active control group and a 6-month follow up measurement, the large sample size of university students at different stages and degrees, and the incorporation of the VR support to facilitate completion to the programme with the possibility of differential analyses. Potential limitations of this study are the voluntary participation of the students, and the utilization of self-report measures exclusively.

DETAILED DESCRIPTION:
Mental health of university students is a noteworthy concern nowadays. Universities are thus challenged to set up effective preventative interventions to help students cope better with university life and improve their mental health. In this regard, it is confirmed that cognitive, behavioral, and mindfulness interventions are effective in reducing symptoms of anxiety in university students.

Mindfulness-based interventions (MBIs) are defined as a type of intervention whose aim is training the mind to adopt a nonjudgmental present-focused awareness. In recent years, these interventions have expanded and have proven to be effective for a variety of clinical and nonclinical populations.This expansion has allowed to study the benefits of mindfulness in university students.

The present study pursue to support this evidence but also to explore the potential benefits of Virtual Reality (VR) around the provision of mindfulness training to university students. VR has showed to be effective for treating several psychological disorders, especially anxiety disorders. However, current research finds promising results when it is incorporated in the third wave of therapy, although the number of studies is still limited yet. A recent study found a high acceptability of VR to practice mindfulness, a significant increase in mindfulness state, and an improved emotional state after one VR mindfulness session.

The main objective of this study is to evaluate the efficacy of a MBI program to reduce stress in university students, in comparison with a relaxation therapy program. The secondary aims are as follows: (1) to analyze the efficacy of a MBI program for improving the psychological well-being and academic functioning of university students, in comparison to the active control group treated with relaxation exercises; (2) to evaluate whether there are differences in the adherence to the mindfulness program, according to the modality in which this mindfulness program has been applied (i.e. with or without VR support); (3) to examine the possible differential effectiveness of each of the sub-groups of mindfulness (i.e. with or without support of the VR) in comparison to the active control group treated with relaxation therapy; (4) to assess the effects of different mindfulness-based VR environments on the emotional and mindfulness states of university students, as well as to evaluate the sensation of immersion caused by each VR environment.

The investigator's main hypothesis is that the provision of mindfulness training will reduce student´s perceived stress of university students in comparison with the university students who have been provided of relaxation training.

This is a randomized, controlled, pragmatic trial, involving three assessment time points (baseline, post-intervention and six-month follow-up). Participants will be randomized into three groups ('mindfulness', 'mindfulness + VR', and 'controls'), considering the secondary objective of evaluating the effectiveness of each mindfulness sub-group separately. Nevertheless, taking into account the primary aim of isolating the common effects of both mindfulness sub-groups, 'mindfulness' and 'mindfulness + VR' will work as an only one group of treatment. 225 participants will be needed: 75 participants in the active control group of relaxation therapy, and 150 participants in the MBI total group. Taking into account all the participants, and assuming a rate of losses of 25%, the total sample has been established in 280 university students.

Several outcomes will be measured and compared between mindfulness (with and without support of VR) and control groups. Three assessment time points will be considered: baseline, post-intervention and six-month follow-up. The investigators will collect data about socio-demographic variables and experience in the use of new technologies, as well as about the primary outcome variable (perceived stress) and secondary outcomes (psychological well-being, academic functioning, mindfulness and compassion).

Socio-demographic data will be described in the baseline by means of frequencies, medians and means, depending on the nature of each of the variables. The treatment conditions will be compared to evaluate the success of randomization by means of Chi-Square test or Fisher test for qualitative variables, Kruskal-Wallis for non-parametric measures and one-way ANOVA for parametric variables. The efficacy of the mindfulness general program compared to the relaxation control group will be analyzed on the main perceived stress variable (PSS), which will be taken continuously. It will be developed by means of a repeated measures design and an intention to treat basis (ITT), using multilevel mixed-effects models,and including time as an independent variable and subjects and presence/absence of VR practices as random effect variables. The efficacy of the general program of mindfulness vs the relaxation control group regarding to psychological well-being, academic functioning, trait mindfulness and self-compassion, will be calculate following the same analytical strategy used for the main analysis. Also the efficacy of the each mindfulness sub-group (with or without VR) vs the control group regarding the main and secondary variables will be estimated - although in this case, the mixed regression model will only include the subjects as a random effects variable.Additionally, possible differences in emotional state, immersion in the VR environment and state mindfulness in the mindfulness + VR sub-group will be explored through each of the VR environments, using the same analytical strategy.

ELIGIBILITY:
Inclusion criteria:

* Students of the Universities of Zaragoza or National Distance Education (UNED), in Spain.
* Being > 18 years of age
* Being in undergraduate or master's degree studies in the referred universities,
* Speaking and writing using the Spanish language and
* Providing written consent form.

Exclusion criteria:

* Suffering a disease which affects the Central Nervous System (CNS),
* Presenting some psychiatric diagnosis or serious psychiatric illness,
* Consumption of drugs or medication that could affect the CNS and
* Having a disorder or illness that may affect their mood.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2018-11-23 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale-10 (PSS) | Baseline
  The Spanish PSS short version provides a reliable and valid measure of perceived stress, with adequate psychometric properties (α = 0.82, test-retest, r = 0.77). Through the PSS, participants are asked to rate on a 5-point Likert-type scale (from 0= "never" to 4= "very often"), how unpredictable, uncontrollable and overloaded have found their life over the past month.
Perceived Stress Scale-10 (PSS) | After programme completion at 6 weeks
  The Spanish PSS short version provides a reliable and valid measure of perceived stress, with adequate psychometric properties (α = 0.82, test-retest, r = 0.77). Through the PSS, participants are asked to rate on a 5-point Likert-type scale (from 0= "never" to 4= "very often"), how unpredictable, uncontrollable and overloaded have found their life over the past month.
Perceived Stress Scale-10 (PSS) | 6-month follow-up
  The Spanish PSS short version provides a reliable and valid measure of perceived stress, with adequate psychometric properties (α = 0.82, test-retest, r = 0.77). Through the PSS, participants are asked to rate on a 5-point Likert-type scale (from 0= "never" to 4= "very often"), how unpredictable, uncontrollable and overloaded have found their life over the past month.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) | Baseline
  This inventory is a widely used, validated measure of anxiety and consists of 20 statements that evaluate how the participants feel at the present moment (State Anxiety), and 20 statements that evaluate how the participants feel in general (Trait anxiety). It uses a 0-3 Likert-type rating scale, being that higher scores are positively correlated with higher levels of anxiety.
State-Trait Anxiety Inventory (STAI) | After programme completion at 6 weeks
  This inventory is a widely used, validated measure of anxiety and consists of 20 statements that evaluate how the participants feel at the present moment (State Anxiety), and 20 statements that evaluate how the participants feel in general (Trait anxiety). It uses a 0-3 Likert-type rating scale, being that higher scores are positively correlated with higher levels of anxiety.
State-Trait Anxiety Inventory (STAI) | 6-month follow-up
  This inventory is a widely used, validated measure of anxiety and consists of 20 statements that evaluate how the participants feel at the present moment (State Anxiety), and 20 statements that evaluate how the participants feel in general (Trait anxiety). It uses a 0-3 Likert-type rating scale, being that higher scores are positively correlated with higher levels of anxiety.
Emotional Regulation Questionnaire (ERQ) | Baseline
  It is a 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal, and (2) Expressive Suppression. The scale consists of 10 items and participants respond using a 7-point Likert scale (from 1 = "strongly disagree", to 7= "strongly agree").
Emotional Regulation Questionnaire (ERQ) | After programme completion at 6 weeks
  It is a 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal, and (2) Expressive Suppression. The scale consists of 10 items and participants respond using a 7-point Likert scale (from 1 = "strongly disagree", to 7= "strongly agree").
Emotional Regulation Questionnaire (ERQ) | 6-month follow-up
  It is a 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal, and (2) Expressive Suppression. The scale consists of 10 items and participants respond using a 7-point Likert scale (from 1 = "strongly disagree", to 7= "strongly agree").
Five Facet Mindfulness Questionnaire (FFMQ) | Baseline
  It is a 39-item self-report measure of mindfulness. The FFMQ is composed of five mindfulness facets: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Respondents indicate on a 5-point Likert scale the degree to which each item is generally true for them, ranging from 1 ("never or very rarely true") to 5 ("very often or always true").
Five Facet Mindfulness Questionnaire (FFMQ) | After programme completion at 6 weeks
  It is a 39-item self-report measure of mindfulness. The FFMQ is composed of five mindfulness facets: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Respondents indicate on a 5-point Likert scale the degree to which each item is generally true for them, ranging from 1 ("never or very rarely true") to 5 ("very often or always true").
Five Facet Mindfulness Questionnaire (FFMQ) | 6-month follow-up
  It is a 39-item self-report measure of mindfulness. The FFMQ is composed of five mindfulness facets: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Respondents indicate on a 5-point Likert scale the degree to which each item is generally true for them, ranging from 1 ("never or very rarely true") to 5 ("very often or always true").
Self-Compassion Scale (SCS) | Baseline
  This scale assesses six facets of behaviours towards self (self-Judgment, self-Kindness, isolation, common humanity, mindfulness, over-identification).The SCS uses a 5-point Likert scale, ranging from 1 ("almost never") to 5 ("almost always").
Self-Compassion Scale (SCS) | After programme completion at 6 weeks
  This scale assesses six facets of behaviours towards self (self-Judgment, self-Kindness, isolation, common humanity, mindfulness, over-identification).The SCS uses a 5-point Likert scale, ranging from 1 ("almost never") to 5 ("almost always").
Self-Compassion Scale (SCS) | 6-month follow-up
  This scale assesses six facets of behaviours towards self (self-Judgment, self-Kindness, isolation, common humanity, mindfulness, over-identification).The SCS uses a 5-point Likert scale, ranging from 1 ("almost never") to 5 ("almost always").
Positive and Negative Affect Schedule (PANAS) | Baseline
  This self-report questionnaire consists of 20 affective descriptors. For each descriptor, respondents rated on a 5-point scale from 1 (very slightly or not at all) to 5 (extremely).
Positive and Negative Affect Schedule (PANAS) | After programme completion at 6 weeks
  This self-report questionnaire consists of 20 affective descriptors. For each descriptor, respondents rated on a 5-point scale from 1 (very slightly or not at all) to 5 (extremely).
Positive and Negative Affect Schedule (PANAS) | 6-month follow-up
  This self-report questionnaire consists of 20 affective descriptors. For each descriptor, respondents rated on a 5-point scale from 1 (very slightly or not at all) to 5 (extremely).
Utrecht Work Engagement Survey Scale-Students (UWES-S) | Baseline
  Consist of 17-item which assess academic engagement. It includes three subscales: vigor (6 items), dedication (5 items), and absorption (6 items). The UWES is scored on a seven-point frequency Likert-type rating scale varying from 0 (never) to 6 (always)
Utrecht Work Engagement Survey Scale-Students (UWES-S) | After programme completion at 6 weeks
  Consist of 17-item which assess academic engagement. It includes three subscales: vigor (6 items), dedication (5 items), and absorption (6 items). The UWES is scored on a seven-point frequency Likert-type rating scale varying from 0 (never) to 6 (always)
Utrecht Work Engagement Survey Scale-Students (UWES-S) | 6-month follow-up
  Consist of 17-item which assess academic engagement. It includes three subscales: vigor (6 items), dedication (5 items), and absorption (6 items). The UWES is scored on a seven-point frequency Likert-type rating scale varying from 0 (never) to 6 (always)
Maslach Burnout Inventory Student Survey (MBI-SS) | Baseline
  It consists of 15 items where the references to work are changed for references to study. This questionnaire includes three subscales: exhaustion (5 items), cynicism (4 items) and (lack of) efficacy (EF; 6 items). Participants have to respond on a Likert-type scale with 7 response options ranged from 0 ("never") to 6 ("always"), and the results are presented in scalar scores.
Maslach Burnout Inventory Student Survey (MBI-SS) | After programme completion at 6 weeks
  It consists of 15 items where the references to work are changed for references to study. This questionnaire includes three subscales: exhaustion (5 items), cynicism (4 items) and (lack of) efficacy (EF; 6 items). Participants have to respond on a Likert-type scale with 7 response options ranged from 0 ("never") to 6 ("always"), and the results are presented in scalar scores.
Maslach Burnout Inventory Student Survey (MBI-SS) | 6-month follow-up
  It consists of 15 items where the references to work are changed for references to study. This questionnaire includes three subscales: exhaustion (5 items), cynicism (4 items) and (lack of) efficacy (EF; 6 items). Participants have to respond on a Likert-type scale with 7 response options ranged from 0 ("never") to 6 ("always"), and the results are presented in scalar scores.
Burnout Clinical Subtype Questionnaire (BCSQ-36) | Baseline
  This scale assesses the three burnout subtypes: frenetic, under-challenged and worn-out. The participants indicate the point to which they agreed with each item using a Likert-type scale with 7 response options ranging from 1 ("never") to 7 ("always").
Burnout Clinical Subtype Questionnaire (BCSQ-36) | After programme completion at 6 weeks
  This scale assesses the three burnout subtypes: frenetic, under-challenged and worn-out. The participants indicate the point to which they agreed with each item using a Likert-type scale with 7 response options ranging from 1 ("never") to 7 ("always").
Burnout Clinical Subtype Questionnaire (BCSQ-36) | 6-month follow-up
  This scale assesses the three burnout subtypes: frenetic, under-challenged and worn-out. The participants indicate the point to which they agreed with each item using a Likert-type scale with 7 response options ranging from 1 ("never") to 7 ("always").
Visual Analog Scale (VAS) | Week 1 (session 1). 5 minutes before starting the Virtual Reality session 1 (baseline)
  This scale assesses the intensity of different emotions before and after the VR intervention. A briefer version of the original measure (16 item emotion) will be used and it will be composed by 7 item emotion (happiness, sadness, anger, surprise, anxiety, relax/calm vigor/energy). Participants can choose responses ranging from 1= "not feeling the emotion at all", to 7 = "feeling the emotion extremely".
Visual Analog Scale (VAS) | Week 1 (session 1). Just after completing the Virtual Reality session 1 (15 minutes from baseline)
  This scale assesses the intensity of different emotions before and after the VR intervention. A briefer version of the original measure (16 item emotion) will be used and it will be composed by 7 item emotion (happiness, sadness, anger, surprise, anxiety, relax/calm vigor/energy). Participants can choose responses ranging from 1= "not feeling the emotion at all", to 7 = "feeling the emotion extremely".
Visual Analog Scale (VAS) | Week 2 (session 2). 5 minutes before starting the Virtual Reality session 2 (baseline)
  This scale assesses the intensity of different emotions before and after the VR intervention. A briefer version of the original measure (16 item emotion) will be used and it will be composed by 7 item emotion (happiness, sadness, anger, surprise, anxiety, relax/calm vigor/energy). Participants can choose responses ranging from 1= "not feeling the emotion at all", to 7 = "feeling the emotion extremely".
Visual Analog Scale (VAS) | Week 2 (session 2). Just after completing the Virtual Reality session 2 (15 minutes from baseline)
  This scale assesses the intensity of different emotions before and after the VR intervention. A briefer version of the original measure (16 item emotion) will be used and it will be composed by 7 item emotion (happiness, sadness, anger, surprise, anxiety, relax/calm vigor/energy). Participants can choose responses ranging from 1= "not feeling the emotion at all", to 7 = "feeling the emotion extremely".
Visual Analog Scale (VAS) | Week 3 (session 3). 5 minutes before starting the Virtual Reality session 3 (baseline)
  This scale assesses the intensity of different emotions before and after the VR intervention. A briefer version of the original measure (16 item emotion) will be used and it will be composed by 7 item emotion (happiness, sadness, anger, surprise, anxiety, relax/calm vigor/energy). Participants can choose responses ranging from 1= "not feeling the emotion at all", to 7 = "feeling the emotion extremely".
Visual Analog Scale (VAS) | Week 3 (session 3). Just after completing the Virtual Reality session 3 (15 minutes from baseline)
  This scale assesses the intensity of different emotions before and after the VR intervention. A briefer version of the original measure (16 item emotion) will be used and it will be composed by 7 item emotion (happiness, sadness, anger, surprise, anxiety, relax/calm vigor/energy). Participants can choose responses ranging from 1= "not feeling the emotion at all", to 7 = "feeling the emotion extremely".
Visual Analog Scale (VAS) | Week 4 (session 4). 5 minutes before starting the Virtual Reality session 4 (baseline)
  This scale assesses the intensity of different emotions before and after the VR intervention. A briefer version of the original measure (16 item emotion) will be used and it will be composed by 7 item emotion (happiness, sadness, anger, surprise, anxiety, relax/calm vigor/energy). Participants can choose responses ranging from 1= "not feeling the emotion at all", to 7 = "feeling the emotion extremely".
Visual Analog Scale (VAS) | Week 4 (session 4). Just after completing the Virtual Reality session 4 (15 minutes from baseline)
  This scale assesses the intensity of different emotions before and after the VR intervention. A briefer version of the original measure (16 item emotion) will be used and it will be composed by 7 item emotion (happiness, sadness, anger, surprise, anxiety, relax/calm vigor/energy). Participants can choose responses ranging from 1= "not feeling the emotion at all", to 7 = "feeling the emotion extremely".
Visual Analog Scale (VAS) | Week 5 (session 5). 5 minutes before starting the Virtual Reality session 5 (baseline)
  This scale assesses the intensity of different emotions before and after the VR intervention. A briefer version of the original measure (16 item emotion) will be used and it will be composed by 7 item emotion (happiness, sadness, anger, surprise, anxiety, relax/calm vigor/energy). Participants can choose responses ranging from 1= "not feeling the emotion at all", to 7 = "feeling the emotion extremely".
Visual Analog Scale (VAS) | Week 5 (session 5). Just after completing the Virtual Reality session 5 (15 minutes from baseline)
  This scale assesses the intensity of different emotions before and after the VR intervention. A briefer version of the original measure (16 item emotion) will be used and it will be composed by 7 item emotion (happiness, sadness, anger, surprise, anxiety, relax/calm vigor/energy). Participants can choose responses ranging from 1= "not feeling the emotion at all", to 7 = "feeling the emotion extremely".
Visual Analog Scale (VAS) | Week 6 (session 6). 5 minutes before starting the Virtual Reality session 6 (baseline)
  This scale assesses the intensity of different emotions before and after the VR intervention. A briefer version of the original measure (16 item emotion) will be used and it will be composed by 7 item emotion (happiness, sadness, anger, surprise, anxiety, relax/calm vigor/energy). Participants can choose responses ranging from 1= "not feeling the emotion at all", to 7 = "feeling the emotion extremely".
Visual Analog Scale (VAS) | Week 6 (session 6). Just after completing the Virtual Reality session 6 (15 minutes from baseline)
  This scale assesses the intensity of different emotions before and after the VR intervention. A briefer version of the original measure (16 item emotion) will be used and it will be composed by 7 item emotion (happiness, sadness, anger, surprise, anxiety, relax/calm vigor/energy). Participants can choose responses ranging from 1= "not feeling the emotion at all", to 7 = "feeling the emotion extremely".
An adaptation (brief version) of the MAAS (Mindful Attention Awareness Scale) (MAAS-State) | Week 1 (session 1). 5 minutes before starting the Virtual Reality session 1 (baseline)
  Each item will be rated on a 7-point Likert-type scale, ranging from 0 ("not at all"), 3 ("somewhat") and 6 ("very much").
An adaptation (brief version) of the MAAS (Mindful Attention Awareness Scale) (MAAS-State) | Week 1 (session 1). Just after completing the Virtual Reality session 1 (15 minutes from baseline)
  Each item will be rated on a 7-point Likert-type scale, ranging from 0 ("not at all"), 3 ("somewhat") and 6 ("very much").
An adaptation (brief version) of the MAAS (Mindful Attention Awareness Scale) (MAAS-State) | Week 2 (session 2). 5 minutes before starting the Virtual Reality session 2 (baseline)
  Each item will be rated on a 7-point Likert-type scale, ranging from 0 ("not at all"), 3 ("somewhat") and 6 ("very much").
An adaptation (brief version) of the MAAS (Mindful Attention Awareness Scale) (MAAS-State) | Week 2 (session 2). Just after completing the Virtual Reality session 2 (15 minutes from baseline)
  Each item will be rated on a 7-point Likert-type scale, ranging from 0 ("not at all"), 3 ("somewhat") and 6 ("very much").
An adaptation (brief version) of the MAAS (Mindful Attention Awareness Scale) (MAAS-State) | Week 3 (session 3). 5 minutes before starting the Virtual Reality session 3 (baseline)
  Each item will be rated on a 7-point Likert-type scale, ranging from 0 ("not at all"), 3 ("somewhat") and 6 ("very much").
An adaptation (brief version) of the MAAS (Mindful Attention Awareness Scale) (MAAS-State) | Week 3 (session 3). Just after completing the Virtual Reality session 3 (15 minutes from baseline)
  Each item will be rated on a 7-point Likert-type scale, ranging from 0 ("not at all"), 3 ("somewhat") and 6 ("very much").
An adaptation (brief version) of the MAAS (Mindful Attention Awareness Scale) (MAAS-State) | Week 4 (session 4). 5 minutes before starting the Virtual Reality session 4 (baseline)
  Each item will be rated on a 7-point Likert-type scale, ranging from 0 ("not at all"), 3 ("somewhat") and 6 ("very much").
An adaptation (brief version) of the MAAS (Mindful Attention Awareness Scale) (MAAS-State) | Week 4 (session 4). Just after completing the Virtual Reality session 4 (15 minutes from baseline)
  Each item will be rated on a 7-point Likert-type scale, ranging from 0 ("not at all"), 3 ("somewhat") and 6 ("very much").
An adaptation (brief version) of the MAAS (Mindful Attention Awareness Scale) (MAAS-State) | Week 5 (session 5). 5 minutes before starting the Virtual Reality session 5 (baseline)
  Each item will be rated on a 7-point Likert-type scale, ranging from 0 ("not at all"), 3 ("somewhat") and 6 ("very much").
An adaptation (brief version) of the MAAS (Mindful Attention Awareness Scale) (MAAS-State) | Week 5 (session 5). Just after completing the Virtual Reality session 5 (15 minutes from baseline)
  Each item will be rated on a 7-point Likert-type scale, ranging from 0 ("not at all"), 3 ("somewhat") and 6 ("very much").
An adaptation (brief version) of the MAAS (Mindful Attention Awareness Scale) (MAAS-State) | Week 6 (session 6). 5 minutes before starting the Virtual Reality session 6 (baseline)
  Each item will be rated on a 7-point Likert-type scale, ranging from 0 ("not at all"), 3 ("somewhat") and 6 ("very much").
An adaptation (brief version) of the MAAS (Mindful Attention Awareness Scale) (MAAS-State) | Week 6 (session 6). Just after completing the Virtual Reality session 6 (15 minutes from baseline)
  Each item will be rated on a 7-point Likert-type scale, ranging from 0 ("not at all"), 3 ("somewhat") and 6 ("very much").
Slater-Usoh-Steed Questionnaire (SUS) | Week 1 (session 1). 5 minutes before starting the Virtual Reality session 1 (baseline)
  Participants response on a 1-7 points Likert scale (1 = "not at all", "at no time" or "something I saw"; 7 = "very much", "almost all of the time" or "some place that I visited") these questions: 1) "Rate your sense of being in the virtual environment"; 2) "To what extent were there times during the experience when the virtual environment was reality for you?"; 3) "To what extent were there times during the experience when the virtual environment became more real or more present for you?";4)"When you think back to the experience, do you think of the virtual environment more as images that you saw or more as some place that you visited?
Slater-Usoh-Steed Questionnaire (SUS) | Week 1 (session 1). Just after completing the Virtual Reality session 1 (15 minutes from baseline)
  Participants response on a 1-7 points Likert scale (1 = "not at all", "at no time" or "something I saw"; 7 = "very much", "almost all of the time" or "some place that I visited") these questions: 1) "Rate your sense of being in the virtual environment"; 2) "To what extent were there times during the experience when the virtual environment was reality for you?"; 3) "To what extent were there times during the experience when the virtual environment became more real or more present for you?";4)"When you think back to the experience, do you think of the virtual environment more as images that you saw or more as some place that you visited?
Slater-Usoh-Steed Questionnaire (SUS) | Week 2 (session 2). 5 minutes before starting the Virtual Reality session 2 (baseline)
  Participants response on a 1-7 points Likert scale (1 = "not at all", "at no time" or "something I saw"; 7 = "very much", "almost all of the time" or "some place that I visited") these questions: 1) "Rate your sense of being in the virtual environment"; 2) "To what extent were there times during the experience when the virtual environment was reality for you?"; 3) "To what extent were there times during the experience when the virtual environment became more real or more present for you?";4)"When you think back to the experience, do you think of the virtual environment more as images that you saw or more as some place that you visited?
Slater-Usoh-Steed Questionnaire (SUS) | Week 2 (session 2). Just after completing the Virtual Reality session 2 (15 minutes from baseline)
  Participants response on a 1-7 points Likert scale (1 = "not at all", "at no time" or "something I saw"; 7 = "very much", "almost all of the time" or "some place that I visited") these questions: 1) "Rate your sense of being in the virtual environment"; 2) "To what extent were there times during the experience when the virtual environment was reality for you?"; 3) "To what extent were there times during the experience when the virtual environment became more real or more present for you?";4)"When you think back to the experience, do you think of the virtual environment more as images that you saw or more as some place that you visited?
Slater-Usoh-Steed Questionnaire" (SUS) | Week 3 (session 3). 5 minutes before starting the Virtual Reality session 3 (baseline)
  Participants response on a 1-7 points Likert scale (1 = "not at all", "at no time" or "something I saw"; 7 = "very much", "almost all of the time" or "some place that I visited") these questions: 1) "Rate your sense of being in the virtual environment"; 2) "To what extent were there times during the experience when the virtual environment was reality for you?"; 3) "To what extent were there times during the experience when the virtual environment became more real or more present for you?";4)"When you think back to the experience, do you think of the virtual environment more as images that you saw or more as some place that you visited?
Slater-Usoh-Steed Questionnaire (SUS) | Week 3 (session 3). Just after completing the Virtual Reality session 3 (15 minutes from baseline)
  Participants response on a 1-7 points Likert scale (1 = "not at all", "at no time" or "something I saw"; 7 = "very much", "almost all of the time" or "some place that I visited") these questions: 1) "Rate your sense of being in the virtual environment"; 2) "To what extent were there times during the experience when the virtual environment was reality for you?"; 3) "To what extent were there times during the experience when the virtual environment became more real or more present for you?";4)"When you think back to the experience, do you think of the virtual environment more as images that you saw or more as some place that you visited?
Slater-Usoh-Steed Questionnaire (SUS) | Week 4 (session 4). 5 minutes before starting the Virtual Reality session 4 (baseline)
  Participants response on a 1-7 points Likert scale (1 = "not at all", "at no time" or "something I saw"; 7 = "very much", "almost all of the time" or "some place that I visited") these questions: 1) "Rate your sense of being in the virtual environment"; 2) "To what extent were there times during the experience when the virtual environment was reality for you?"; 3) "To what extent were there times during the experience when the virtual environment became more real or more present for you?";4)"When you think back to the experience, do you think of the virtual environment more as images that you saw or more as some place that you visited?
Slater-Usoh-Steed Questionnaire (SUS) | Week 4 (session 4). Just after completing the Virtual Reality session 4 (15 minutes from baseline)
  Participants response on a 1-7 points Likert scale (1 = "not at all", "at no time" or "something I saw"; 7 = "very much", "almost all of the time" or "some place that I visited") these questions: 1) "Rate your sense of being in the virtual environment"; 2) "To what extent were there times during the experience when the virtual environment was reality for you?"; 3) "To what extent were there times during the experience when the virtual environment became more real or more present for you?";4)"When you think back to the experience, do you think of the virtual environment more as images that you saw or more as some place that you visited?
Slater-Usoh-Steed Questionnaire (SUS) | Week 5 (session 5). 5 minutes before starting the Virtual Reality session 5 (baseline)
  Participants response on a 1-7 points Likert scale (1 = "not at all", "at no time" or "something I saw"; 7 = "very much", "almost all of the time" or "some place that I visited") these questions: 1) "Rate your sense of being in the virtual environment"; 2) "To what extent were there times during the experience when the virtual environment was reality for you?"; 3) "To what extent were there times during the experience when the virtual environment became more real or more present for you?";4)"When you think back to the experience, do you think of the virtual environment more as images that you saw or more as some place that you visited?
Slater-Usoh-Steed Questionnaire (SUS) | Week 5 (session 5). Just after completing the Virtual Reality session 5 (15 minutes from baseline)
  Participants response on a 1-7 points Likert scale (1 = "not at all", "at no time" or "something I saw"; 7 = "very much", "almost all of the time" or "some place that I visited") these questions: 1) "Rate your sense of being in the virtual environment"; 2) "To what extent were there times during the experience when the virtual environment was reality for you?"; 3) "To what extent were there times during the experience when the virtual environment became more real or more present for you?";4)"When you think back to the experience, do you think of the virtual environment more as images that you saw or more as some place that you visited?
Slater-Usoh-Steed Questionnaire (SUS) | Week 6 (session 6). 5 minutes before starting the Virtual Reality session 6 (baseline)
  Participants response on a 1-7 points Likert scale (1 = "not at all", "at no time" or "something I saw"; 7 = "very much", "almost all of the time" or "some place that I visited") these questions: 1) "Rate your sense of being in the virtual environment"; 2) "To what extent were there times during the experience when the virtual environment was reality for you?"; 3) "To what extent were there times during the experience when the virtual environment became more real or more present for you?";4)"When you think back to the experience, do you think of the virtual environment more as images that you saw or more as some place that you visited?
Slater-Usoh-Steed Questionnaire (SUS) | Week 6 (session 6). Just after completing the Virtual Reality session 6 (15 minutes from baseline)
  Participants response on a 1-7 points Likert scale (1 = "not at all", "at no time" or "something I saw"; 7 = "very much", "almost all of the time" or "some place that I visited") these questions: 1) "Rate your sense of being in the virtual environment"; 2) "To what extent were there times during the experience when the virtual environment was reality for you?"; 3) "To what extent were there times during the experience when the virtual environment became more real or more present for you?";4)"When you think back to the experience, do you think of the virtual environment more as images that you saw or more as some place that you visited?

CONTACTS AND LOCATIONS:
Overall Officials: Javier García-Campayo, phD, Principal Investigator — Miguel Servet University Hospital, Zaragoza, Spain
Locations (1):
- Department of Psychiatry. Miguel Servet University Hospital, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes
Databases will be shared for replication studies upon request and reasonable conditions.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be shared when the study will be published. Length: 5 years.
Access Criteria: Upon request and reasonable conditions.

REFERENCES:
- [Background] Neff, K. D. Development and validation of a scale to measure self-compassion. Self and Identity, 2, 223-250, 2003.
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] S. Cohen, G. Williamson, Perceived stress in a probability sample of the United States, in: S. Spacapan, S. Oskamp (Eds.), The Social Psychology of Health, Sage, Newbury Park, CA, 1988.
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Schaufeli, W. B., Salanova, M., Gonzàlez-Romá, V., & Bakker, A. B. (2002). The measurement of engagement and burnout: A two sample confirmatory factor analytic approach. Journal of Happiness Studies, 3, 71-92. doi:10.1023/A:1015630930326
- [Background] Schaufeli WB, Martínez I, Marqués-Pinto A, Salanova M, Bakker A: Burnout and engagement in university students: A cross-national study. Journal of Cross-Cultural Studies. 2002, 33: 464-481.
- [Background] Gross JJ, Levenson RW. Emotion elicitation using films. Cogn Emot. 1995 Jan; 9(1):87-108.
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Slater M, Usoh M, Steed A. Depth of Presence in Virtual Environments. Presence Teleoperators Virtual Environ. 1994 Jan; 3(2):130-44.
- [Background] Navarro-Haro MV, Lopez-Del-Hoyo Y, Campos D, Linehan MM, Hoffman HG, Garcia-Palacios A, Modrego-Alarcon M, Borao L, Garcia-Campayo J. Meditation experts try Virtual Reality Mindfulness: A pilot study evaluation of the feasibility and acceptability of Virtual Reality to facilitate mindfulness practice in people attending a Mindfulness conference. PLoS One. 2017 Nov 22;12(11):e0187777. doi: 10.1371/journal.pone.0187777. eCollection 2017. PMID 29166665
- [Background] Regehr C, Glancy D, Pitts A. Interventions to reduce stress in university students: a review and meta-analysis. J Affect Disord. 2013 May 15;148(1):1-11. doi: 10.1016/j.jad.2012.11.026. Epub 2012 Dec 13. PMID 23246209
- [Background] Conley CS, Shapiro JB, Kirsch AC, Durlak JA. A meta-analysis of indicated mental health prevention programs for at-risk higher education students. J Couns Psychol. 2017 Mar;64(2):121-140. doi: 10.1037/cou0000190. PMID 28277730
- [Background] Gotink RA, Chu P, Busschbach JJ, Benson H, Fricchione GL, Hunink MG. Standardised mindfulness-based interventions in healthcare: an overview of systematic reviews and meta-analyses of RCTs. PLoS One. 2015 Apr 16;10(4):e0124344. doi: 10.1371/journal.pone.0124344. eCollection 2015. PMID 25881019 (Retraction: PMID 30978236 PLoS One. 2019 Apr 12;14(4):e0215608)
- [Background] Khoury B, Lecomte T, Fortin G, Masse M, Therien P, Bouchard V, Chapleau MA, Paquin K, Hofmann SG. Mindfulness-based therapy: a comprehensive meta-analysis. Clin Psychol Rev. 2013 Aug;33(6):763-71. doi: 10.1016/j.cpr.2013.05.005. Epub 2013 Jun 7. PMID 23796855
- [Background] Montero-Marin J, Garcia-Campayo J. A newer and broader definition of burnout: validation of the "Burnout Clinical Subtype Questionnaire (BCSQ-36)". BMC Public Health. 2010 Jun 2;10:302. doi: 10.1186/1471-2458-10-302. PMID 20525178
- [Derived] Modrego-Alarcon M, Lopez-Del-Hoyo Y, Garcia-Campayo J, Perez-Aranda A, Navarro-Gil M, Beltran-Ruiz M, Morillo H, Delgado-Suarez I, Olivan-Arevalo R, Montero-Marin J. Efficacy of a mindfulness-based programme with and without virtual reality support to reduce stress in university students: A randomized controlled trial. Behav Res Ther. 2021 Jul;142:103866. doi: 10.1016/j.brat.2021.103866. Epub 2021 Apr 26. PMID 33957506